CLINICAL TRIAL: NCT06859164
Title: Genicular Artery Embolization for Reducing Pain in Symptomatic Knee Osteoarthritis: A Pilot Randomized Sham-Controlled Study
Brief Title: Genicular Artery Embolization for Reducing Pain in Medically Refractory Symptomatic Knee Osteoarthritis
Acronym: SHAM-PAIN
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB24-1674; 1R21AR082123-01A1 (NIH)
Record Dates: First submitted 2025-02-23; First posted 2025-03-05 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Knee Osteoarthritis; Knee Osteoarthritis (Knee OA); Knee Osteoarthritis (OA)
Keywords: Osteoarthritis; Knee pain; MSK pain; Musculoskeletal Pain; Osteoarthritis of the knee; GAE; Genicular artery embolization; Geniculate artery embolization; MSK embolization; Musculoskeletal Embolization; Embolization; Musculoskeletal; Temporary Embolization
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis; Musculoskeletal Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- GAE Arm (Experimental): In this study, GAE is performed using the Lipiojoint technique described by Sapoval et al. This method utilizes a 3:1 emulsion of Lipiodol® (a transient embolic agent that penetrates distally to about 30 microns) and Optiray® to target the genicular arteries supplying areas of synovial hypervascularity and neo-angiogenesis. The embolic effect is temporary-lasting roughly 10 minutes-after which angiographic imaging shows resolution of the embolization with no damage to the surrounding skin, tendon, or bone. The endpoint of the procedure is to achieve complete stasis in the targeted vessels. 20 participants will be randomly allocated to this arm.
  Interventions: Procedure: Genicular Artery Embolization; Device: Lipiodol; Procedure: Simple angiogram
- Sham Arm (Sham Comparator): Participants assigned to the sham group undergo a similar preparatory process, including angiography and catheterization of all genicular arteries. However, no embolic agent is administered. Instead, after performing selective angiograms, these participants do not receive any embolization. 20 participants will be randomly allocated to this arm.
  Interventions: Procedure: Simple angiogram

INTERVENTIONS:
Procedure: Genicular Artery Embolization — Embolization of genicular arteries that demonstrate neoangiogenesis or blush on angiogram.
  Other Names: GAE; Geniculate Artery Embolization
  Arms: GAE Arm
Device: Lipiodol — 3:1 emulsion of Lipiodol to Optiray
  Arms: GAE Arm
Procedure: Simple angiogram — Simple angiogram of the genicular arteries

SUMMARY:
Genicular Artery Embolization for Reducing Pain in Symptomatic Knee Osteoarthritis: A Pilot Randomized Sham-Controlled Study (SHAM-PAIN) is a NIH-NIAMS funded project designed to assess enrollment feasibility and detect any differences between GAE and a similar sham intervention in reducing KOA-related pain at 3 months as measured by the Knee injury and Osteoarthritis Outcome Score (KOOS) pain subscore. Additionally, this study aims to determine the magnitude of difference in pain response between GAE and sham to adequately power a larger, more definitive randomized sham-controlled trial (RCT). The influence of psychosocial and psychocognitive factors, changes in analgesic use, and conditions of knee joint cartilage and effusion will similarly be explored to determine their impacts on perceived pain response to GAE.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 40-80
* Bilateral or unilateral knee pain attributed to osteoarthritis (treat the knee with greater pain-if equal, patient chooses)
* Grade 2-4 osteoarthritis on standing weight-bearing knee radiographs per the Kellgren-Lawrence grading scale
* Knee pain > 6 months, refractory to conservative non-operative management, and scored ≥ 4 on Visual Analog Scale (VAS) (e.g., rest, activity modification, weight control, bracing, supervised physical therapy, nonsteroidal anti-inflammatory drugs (NSAIDs), acetaminophen, oral opiates, intra-articular hyaluronic acid, PRP, stem cells, and/or oral/injectable corticosteroids)
* Refusal of intra-articular corticosteroid injection

Exclusion Criteria:

* Active malignancy
* Active infection of the affected knee
* Corticosteroid injection of the affected knee within 3 months of enrollment
* Rheumatoid arthritis or other seronegative arthropathy
* Previous surgery of the affected knee (e.g., meniscus repair, meniscectomy, anterior cruciate ligament (ACL)/posterior cruciate ligament (PCL) reconstruction, chondroplasty, microfracture, loose-body removal, synovectomy, lateral release, patellar/quadriceps tendon repair, total or partial knee replacement, osteotomy, cartilage transplant), except diagnostic arthroscopy
* Grade 0-1 osteoarthritis per Kellgren-Lawrence grading scale of the affected knee
* Pregnancy or expected pregnancy
* GFR < 60 mL/min/1.73 m²
* Anaphylactic reaction to iodinated contrast
* Moderate to severe pain in other ipsilateral lower-limb joints (ankle, hip) with VAS > 4
* Body weight > 400 lbs (unsafe for angiography)
* Peripheral arterial disease of the treated extremity (Rutherford Grade 2 or greater)
* Type 1 diabetes mellitus
* Long-acting corticosteroid use within 6 months (3 months for short-acting)
* History or other evidence of acute kidney injury (AKI)
* History of reaction to contrast media, bronchial asthma, or allergic disorders
* History of hypersensitivity to gadolinium-based contrast agents (GBCAs)
* Chronic widespread generalized pain >4 on VAS pain scale, including neuropathic pain
* Major depressive disorder within 2 years before screening
* Other severe psychiatric disorder (e.g., schizophrenia, bipolar disorder)
* Suicide attempt or suicidal behavior within 30 days before screening
* Diagnosis of fibromyalgia
* Considering total knee replacement in the next year
* Any other condition, unwillingness, or inability that, in the investigator's opinion, could jeopardize the subject's safety or protocol compliance

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Reduction in KOOS pain subscore | 3 months
  Percent change in KOOS pain subscale score, scaled to a range of 0-100, from baseline to 3 months post-randomization of both GAE and sham groups.

SECONDARY OUTCOMES:
WOMAC knee pain and dysfunction | 1, 3, 6, 9, and 12 months.
  Reduction in knee pain and dysfunction (WOMAC) at 1, 3, 6, 9, and 12 months.
KOOS pain and dysfunction | 1, 3, 6, 9, and 12 months
  Absolute reduction in knee pain and dysfunction (KOOS) at 1, 3, 6, 9, and 12 months
VAS Score | 0, 1, 6, 9, and 12 months
  Visual Analog Score (VAS) for pain at 0, 1, 6, 9, and 12 months post treatment
Crossover | 3 months
  Rate of cross-over from sham to GAE at 3 months
Analgesic Reduction | Baseline, 1, 3, 6, 9, and 12 months post intervention
  Usage of opiate/analgesic medications at baseline, 1, 3, 6, 9, and 12 months post intervention
Whole Knee Synovitis Scoring | Baseline and 3 months
  Contrast Enhanced MRI with Whole Knee Synovitis Scoring at baseline and 3 months
Perfusion | Procedure
  Perfusion quantification using pre and post embolization using CT-Perfusion scanning
Knee replacement | 3 months
  Rate of total knee replacement at 3 months
Corticosteroid injection usage | Baseline, 1, 3, 6, 9, and 12 months post intervention
  Corticosteroid injection rate usage at baseline, 1, 3, 6, 9, and 12 months post intervention

CONTACTS AND LOCATIONS:
Overall Officials: Osman Ahmed, MD, Principal Investigator — University of Chicago Department of Radiology
Locations (1):
- University of Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided
Will need to be considered on an individual basis given the desire to protect PHI

REFERENCES:
- [Background] Ahmed O, Block J, Mautner K, Plancher K, Anitescu M, Isaacson A, Filippiadis DK, Epelboym Y, Bercu Z, Mitchell JW, Cristescu M, White SB, Prologo JD. Percutaneous Management of Osteoarthritis in the Knee: Proceedings from the Society of Interventional Radiology Research Consensus Panel. J Vasc Interv Radiol. 2021 Jun;32(6):919.e1-919.e6. doi: 10.1016/j.jvir.2021.03.409. Epub 2021 Mar 6. No abstract available. PMID 33689834
- [Background] Ahmed O, Epelboym Y, Haskal ZJ, Okuno Y, Taslakian B, Sapoval M, Nikolic B, Golzarian J, Gaba RC, Little M, Isaacson A, Padia SA, Sze DY. Society of Interventional Radiology Research Reporting Standards for Genicular Artery Embolization. J Vasc Interv Radiol. 2024 Aug;35(8):1097-1103. doi: 10.1016/j.jvir.2024.04.018. Epub 2024 Apr 27. PMID 38685470
- [Background] Dariushnia SR, Redstone EA, Heran MKS, Cramer HR Jr, Ganguli S, Gomes AS, Hogan MJ, Himes EA, Patel S, Schiro BJ, Lewis CA. Society of Interventional Radiology Quality Improvement Standards for Percutaneous Transcatheter Embolization. J Vasc Interv Radiol. 2021 Mar;32(3):476.e1-476.e33. doi: 10.1016/j.jvir.2020.10.022. No abstract available. PMID 33640083
- [Background] Parry E, Ogollah R, Peat G. Significant pain variability in persons with, or at high risk of, knee osteoarthritis: preliminary investigation based on secondary analysis of cohort data. BMC Musculoskelet Disord. 2017 Feb 14;18(1):80. doi: 10.1186/s12891-017-1434-3. PMID 28196504
- [Background] Derkach M, Al Sayah F, Ohinmaa A, Svenson LW, Johnson JA. Comparative performance of the EuroQol EQ-5D-5L and the CDC healthy days measures in assessing population health. J Patient Rep Outcomes. 2022 Jun 13;6(1):64. doi: 10.1186/s41687-022-00474-7. PMID 35696002
- [Background] Binkley JM, Stratford PW, Lott SA, Riddle DL. The Lower Extremity Functional Scale (LEFS): scale development, measurement properties, and clinical application. North American Orthopaedic Rehabilitation Research Network. Phys Ther. 1999 Apr;79(4):371-83. PMID 10201543
- [Background] Salaffi F, Leardini G, Canesi B, Mannoni A, Fioravanti A, Caporali R, Lapadula G, Punzi L; GOnorthrosis and Quality Of Life Assessment (GOQOLA). Reliability and validity of the Western Ontario and McMaster Universities (WOMAC) Osteoarthritis Index in Italian patients with osteoarthritis of the knee. Osteoarthritis Cartilage. 2003 Aug;11(8):551-60. doi: 10.1016/s1063-4584(03)00089-x. PMID 12880577
- [Background] Little MW, O'Grady A, Briggs J, Gibson M, Speirs A, Al-Rekabi A, Yoong P, Ariyanayagam T, Davies N, Tayton E, Tavares S, MacGill S, McLaren C, Harrison R. Genicular Artery embolisation in Patients with Osteoarthritis of the Knee (GENESIS) Using Permanent Microspheres: Long-Term Results. Cardiovasc Intervent Radiol. 2024 Dec;47(12):1750-1762. doi: 10.1007/s00270-024-03752-7. Epub 2024 May 31. PMID 38819473
- [Background] Padia SA, Genshaft S, Blumstein G, Plotnik A, Kim GHJ, Gilbert SJ, Lauko K, Stavrakis AI. Genicular Artery Embolization for the Treatment of Symptomatic Knee Osteoarthritis. JB JS Open Access. 2021 Oct 21;6(4):e21.00085. doi: 10.2106/JBJS.OA.21.00085. eCollection 2021 Oct-Dec. PMID 34703964
- [Background] Sapoval M, Querub C, Pereira H, Pellerin O, Boeken T, Di Gaeta A, Ahmar MA, Lefevre-Colau MM, Nguyen C, Daste C, Lacroix M, Laredo JD, Sabatier B, Martelli N, Chatellier G, Dean C, Rannou F. Genicular artery embolization for knee osteoarthritis: Results of the LipioJoint-1 trial. Diagn Interv Imaging. 2024 Apr;105(4):144-150. doi: 10.1016/j.diii.2023.12.003. Epub 2023 Dec 14. PMID 38102013
- [Background] Lim WB, Al-Dadah O. Conservative treatment of knee osteoarthritis: A review of the literature. World J Orthop. 2022 Mar 18;13(3):212-229. doi: 10.5312/wjo.v13.i3.212. eCollection 2022 Mar 18. PMID 35317254
- [Background] Heidari B. Knee osteoarthritis prevalence, risk factors, pathogenesis and features: Part I. Caspian J Intern Med. 2011 Spring;2(2):205-12. PMID 24024017
- [Background] GBD 2021 Osteoarthritis Collaborators. Global, regional, and national burden of osteoarthritis, 1990-2020 and projections to 2050: a systematic analysis for the Global Burden of Disease Study 2021. Lancet Rheumatol. 2023 Aug 21;5(9):e508-e522. doi: 10.1016/S2665-9913(23)00163-7. eCollection 2023 Sep. PMID 37675071